CLINICAL TRIAL: NCT02044068
Title: Prevention of Hepatitis B Virus Mother-to-Child Transmission (MTCT) From HIV-HBV Co-infected Pregnant Women by Use of Nucleosides/Nucleotides Analogues With Dual Activity During Pregnancy.
Brief Title: Hepatitis B Virus Vertical Transmission From HIV-HBV Co-infected Women
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, Professor at Paris VII Denis Diderot University, physician, Hopital Lariboisière
Other Study IDs: Liver003
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Vertical Disease Transmission; HBV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children born from HIV-HBV women: Studying retrospectively their status for HBs Ag and HBc Ab

SUMMARY:
Vertical HIV transmission has been dramatically reduced by the use of combined antiretroviral therapy in HIV-infected pregnant women. Among the most often used drugs, several have dual activity, against HIV and HBV: lamivudine, emtricitabine, tenofovir. Studies about vertical HBV transmission from HIV-HBV co-infected pregnant women are rare in developed countries. The study hypothesis is a major reduction of the risk of HBV vertical transmission.

DETAILED DESCRIPTION:
Mother-to-Child HIV transmission has been dramatically reduced by the use of combined antiretroviral therapy in HIV-infected pregnant women, both in developed and in developing countries. Among the most often used drugs, several have dual activity, against HIV and HBV: lamivudine, emtricitabine, tenofovir; they can be used as a combo, as tenofovir+emtricitabine for instance. Studies about vertical HBV transmission from HIV-HBV co-infected pregnant women are rare in developed countries. The study hypothesis is a major reduction of the risk of HBV vertical transmission in this context, justifying this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* children born in the Maternity Department from HIV-HBV co-infected women
* whose mother was given a treatment with dual activity (HIV and HBV) during pregnancy

Exclusion Criteria:

* no

Ages: 9 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children born in the Maternity Department, Lariboisiere Hospital, Paris, France, from HIV-HBV co-infected women
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hepatitis B sAg status in children born from HIV-Hepatitis B Virus co-infected women | up to 10 years (expected average: 5 years)

SECONDARY OUTCOMES:
Antibodies (Ab) against Hepatitis B core antigen in children | up to 10 years (expected average: 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O SELLIER, MD, PhD, Principal Investigator — Hopital Lariboisiere, Paris, France
Locations (1):
- Hopital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sellier PO, Schnepf N, Amarsy R, Maylin S, Lopes A, Mazeron MC, Flateau C, Morgand M, Ciraru-Vigneron N, Berthe A, Simoneau G, Evans J, Souak S, Matheron S, Benifla JL, Simon F, Bergmann JF. Short article: Hepatitis B virus status in children born to HIV/HBV coinfected women in a French hospital: a cross-sectional study. Eur J Gastroenterol Hepatol. 2016 Mar;28(3):328-32. doi: 10.1097/MEG.0000000000000559. PMID 26709883